CLINICAL TRIAL: NCT00723840
Title: Assessment of the Social Cost of Crohn's Disease (COsto Sociale Della Malattia di CrOhn - COSMO): Economic and Quality of Life Aspects
Brief Title: Assessment of the Social Cost of Crohn's Disease: Economic and Quality of Life Aspects (Study P04560)
Acronym: COSMO
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: P04560
Record Dates: First submitted 2008-07-25; First posted 2008-07-29 (Estimated); Results first posted 2011-04-29 (Estimated); Last update posted 2015-07-30 (Estimated); Status verified 2015-07

CONDITIONS: Inflammatory Bowel Disease; Crohn's Disease
Keywords: EuroQOL (EQ-5D)
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Crohn's Disease Participants: Participants with Crohn's Disease for at least 6 months, who have a Crohn's Disease Activity Index (CDAI) score >= 150. The CDAI score evaluates Crohn's disease symptoms - a score of 150 or below indicates remission and a score above 450 indicates extremely severe disease.
  These participants have active disease despite drug therapy.
  Interventions: Other: Observational Studies: participants treated according to the real clinical practice.

INTERVENTIONS:
Other: Observational Studies: participants treated according to the real clinical practice. — No intervention was administered to the participants specifically for the purpose this study. Participant could be on any drug therapy.
  Other Names: Crohn's Disease Participants

SUMMARY:
This observational study will evaluate the social cost and quality of life of participants who have had Crohn's Disease for at least 6 months and have active disease despite drug therapy. Participants are followed for a total of 18 months.

DETAILED DESCRIPTION:
Participants for this study will be enrolled from 25 gastroenterology sites, even spread across Italy. Each center will enroll between 10 and 40 participants each.

ELIGIBILITY:
Inclusion Criteria:

* participant must:

  * be between 18 and 70 years of age,
  * have active Crohn's disease (CD) with CDAI score >= 150 (as per amended protocol) in spite of drug therapy, or active fistulizing disease,
  * be diagnosed with CD for at least 6 months,
  * sign the informed consent,
  * be capable of understanding the study and replying to the questionnaires.

Exclusion Criteria:

* Participants who are unreliable in filling out questionnaires,
* Participants with diseases which may interfere with the cost's of CD or its complications,
* Participants who are participating in a clinical trial

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Crohn's Disease for at least 6 months who have active disease despite drug therapy and are seen at one of 25 gastroenterology centers spread across Italy.
Sampling Method: Non-Probability Sample
Enrollment: 245 (Actual)
Dates: Start 2006-09; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

REFERENCES:
- [Result] Benedini V, Caporaso N, Corazza GR, Rossi Z, Fornaciari G, Cottone M, Frosini G, Caruggi M, Ottolini C, Colombo GL. Burden of Crohn's disease: economics and quality of life aspects in Italy. Clinicoecon Outcomes Res. 2012;4:209-18. doi: 10.2147/CEOR.S31114. Epub 2012 Jul 24. PMID 22866007

RESULTS

PARTICIPANT FLOW:
Groups:
- Crohn's Disease Participants: Participants with Crohn's Disease for at least 6
  months, who have a Crohn's Disease Activity Index
  (CDAI) score >= 150, seen at one of 25 gastroenterology centers spread across Italy. The CDAI score evaluates Crohn's disease symptoms - a score of 150 or below
  indicates remission and a score above 450 indicates extremely severe disease.
Period: Overall Study
Arm/Group | Crohn's Disease Participants
Started | 245
Completed | 163
Not Completed | 82
Not completed — Lost to Follow-up | 2
Not completed — Failure to return | 18
Not completed — Withdrawal by Subject | 55
Not completed — Serious Adverse Events | 3
Not completed — Other Medical Event | 2
Not completed — Unspecified reason | 2

BASELINE CHARACTERISTICS:
Arm/Group | Crohn's Disease Participants
Number analyzed (Participants) | 162
Age, Customized [Number; unit: participants] — Baseline characteristics for participants included in the pharmacoeconomic analysis. Of the enrolled population, a total of 82 subjects interrupted the study prematurely. In addition, for one participant, the age and sex were not available. These participants were not included in the pharmacoeconomic analysis. Therefore, the number of participants analyzed for this study is 162.
  participants
    <18 years | 0
    Between 18 and 34 years | 46
    Between 35 and 44 years | 43
    Between 45 and 64 years | 61
    >=65 years | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81
  Male | 81
Region of Enrollment [Number; unit: participants]
  Italy | 162

OUTCOME MEASURES:

1. Primary Outcome: Cost of Illness in Participants With Crohn's Disease
Description: Direct health care costs, non health care costs and costs for productivity loss were calculated by observation period in Crohn's Disease participants (in active phase) with a CDAI score >= 150.
  Direct health care costs refer to the resources used to prevent and treat a disease. Indirect costs include expenses for a participant's (or their caregiver's) transport, home assistance or home nursing assistance. Costs for productivity loss include the participant's (or their caregiver's) productivity loss or time loss.
Time Frame: Baseline, 6, 12, and 18 months
Population: Of the enrolled population, a total of 82 subjects interrupted the study prematurely. For one participant, the age and sex were not available. These participants were not included in the pharmacoeconomic analysis.
Measure: Number; unit: Euros
Groups:
- Baseline: Costs per participant at baseline in Euros
- 6 Months: Costs per participant at 6 months in Euros
- 12 Months: Costs per participant at 12 months in Euros
- 18 Months: Costs per participant at 18 months in Euros
Arm/Group | Baseline | 6 Months | 12 Months | 18 Months
Number analyzed (Participants) | 162 | 154 | 154 | 155
Euros
  Health care direct costs | 6088.40 | 6169.62 | 5594.00 | 5825.80
  Non-health care costs | 1132.60 | 348.70 | 143.10 | 173.60
  Costs for productivity loss | 2173.00 | 1455.50 | 1199.10 | 740.20

2. Primary Outcome: EuroQoL (Quality of Life)-5 Dimensions (EQ-5D) Scores in Participants With Crohn's Disease
Description: EQ-5D was calculated for the pharmacoeconomics analysis to evaluate quality of life (QoL) in participants in the active phase with Crohn's Disease and had a CDAI score >= 150.
  EQ-5D is a participant answered questionnaire scoring 5 dimensions - mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The EQ-5D total score ranges from 0 (worst health state) to 1 (perfect health state) and 1 reflects the best outcome.
Time Frame: Baseline, 6, 12, and 18 months
Population: as for outcome 1
Measure: Number; unit: Score on a scale
Groups:
- Baseline: QoL scores per participant at baseline
- 6 Months: QoL scores per participant at 6 months
- 12 Months: QoL scores per participant at 12 months
- 18 Months: QoL scores per participant at 18 months
Arm/Group | Baseline | 6 Months | 12 Months | 18 Months
Number analyzed (Participants) | 162 | 154 | 154 | 155
Score on a scale | 0.558 | 0.682 | 0.728 | 0.739

ADVERSE EVENTS:
Arm/Group | Crohn's Disease Participants
Serious Adverse Events (participants affected / at risk) | 3/245
Other Adverse Events (participants affected / at risk) | 0/245
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Crohn's Disease Participants (N=245)
Intestinal stenosis (Gastrointestinal disorders) | 1 (1)
Drug ineffective (General disorders) | 1 (1)
Abdominal abscess (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The disclosure restriction on the principal investigator (PI) is that the PI agrees not to publish or publicly present any results of the study without the prior written permission of the sponsor. The PI further agrees to allow the sponsor to review, 30 days prior to submission for publication or presentation, copies of abstracts or manuscripts for publication (including texts of oral presentations) which report any results of the study.